CLINICAL TRIAL: NCT03916718
Title: The Dementia Care EcoSystem: The Feasibility of a Care Management Program Addressing Healthcare Quality, Access, and Cost for Patients With Dementia and Their Caregivers
Brief Title: Care EcoSystem: Ochsner Health System
Status: Completed | Type: Observational
Sponsor: Ochsner Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 2018241
Record Dates: First submitted 2019-04-10; First posted 2019-04-16 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2021-02

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dementia: The target population includes patients seen at Ochsner Clinic Foundation, >=55 years old, diagnosed with dementia, and meeting other inclusion/exclusion criteria. this study will recruit subjects identified as high utilizers of the Ochsner System. This will be defined by >= 2 ED visits, >= 2 Hospitalizations, or some combination prior to baseline. We will co-variate by insurance plan.
  Interventions: Behavioral: Care EcoSystem

INTERVENTIONS:
Behavioral: Care EcoSystem — This is a care management program and health care outcomes feasibility study utilizing the dementia Care Ecosystem (CE) program developed at UCSF and tailored to high need Ochsner PWD (patient with dementia) and their CGs (caregivers). Dyads (CGs and PWD) will receive a tailored clinical assessment addressing dementia severity, PWD and CG needs, education/strategies to management common dementia issues, medical issues and medication reconciliation, caregiver wellness strategies, linkages to community-based resources, advance care planning, education about the risk of ED and hospitalization, and care coordination with other specialties. Dyads will be followed on a monthly basis to monitor needs, provide support, and problem solve issues.

SUMMARY:
1. To determine the feasibility and acceptability of the Care Ecosystem program in the Ochsner clinical setting.
2. To assess the effect of the Care Ecosystem program on health care cost and quality care quality as measured by primary outcome variables.

   * Adapted from the Care Ecosystem, memory.ucsf.edu/Care-Ecosystem

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥55 years of age at baseline
* Probable dementia diagnosis as evidenced by one or more of the following criteria:

  * Dementia listed on medical record problem list as of January 1, 2015 or later, or, in the opinion of the referring provider has dementia
  * Prescribed with any of the following: donepezil, memantine, galantamine HBR, rivastigmine, or tartrate; or, in the opinion of the referring provider, could take such medication
* Lives in community

Exclusion Criteria:

* Documented history of Multiple Sclerosis, ALS, Traumatic Brain Injury, Huntington's Disease, Schizophrenia, Bipolar Disorder, or current Substance Abuse Disorder
* Lives in a nursing home or assisted living facility
* Unable to complete monthly telehealth or phone visits

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population includes patients seen at Ochsner Clinic Foundation, >=55 years old, diagnosed with dementia, and meeting other inclusion/exclusion criteria. this study will recruit subjects identified as high utilizers of the Ochsner System. This will be defined by >= 2 ED visits, >= 2 Hospitalizations, or some combination prior to baseline. We will co-variate by insurance plan.
Sampling Method: Non-Probability Sample
Enrollment: 290 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Rate of ED and Hospital Admissions | through study completion, an average of 1 year
  Cost
Quick Dementia Rating Scale (QDRS) | through study completion, an average of 1 year
  Construct: Dementia severity Sum total score Normal 0-1 Mild cognitive impairment 2-5 Mild dementia 6-12 Moderate dementia 13-20 Severe dementia 20-30
Quality of Life in Dementia (QUALI-DEM) | through study completion, an average of 1 year
  Construct: Dementia patient quality of life Subscales Care Relationship (0-9) Positive Affect (0-12) Negative Affect (0-6) Restless Tense Behavior (0-9) Social Relations (0-9) Social Isolation (0-9)
  Higher scores= more of that behavior
Zarit Caregiver Burden Scale- Short Form | through study completion, an average of 1 year
  Construct: Family/Caregiver quality of life Sum total score 0-48, higher scores indicate more burden

SECONDARY OUTCOMES:
Rate of Falls | through study completion, an average of 1 year
Rate of UTIs | through study completion, an average of 1 year
Rate of medication change | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: R. John Sawyer, PhD, Principal Investigator — Ochsner Health System
Locations (1):
- Ochsner Health System, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: UCSF Care Ecosystem — https://memory.ucsf.edu/care-ecosystem